CLINICAL TRIAL: NCT03350009
Title: Markers in Follicular Fluid and in Embryo Culture Medium as a Marker of Oocyte and Embryo Quality
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CMC-16-0163-CTIL
Record Dates: First submitted 2017-11-02; First posted 2017-11-22 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Infertility/Sterility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High and low grade embryos: The distribution for the high and low grade embryos is based on common morphological grading criteria.
- High and low quality follicles: The distribution for the high and low grade oocytes is based on common morphological grading criteria and on different features of the participants such as age.

SUMMARY:
Assessment of the quality of follicular fluid and early embryo via chemical markers.

DETAILED DESCRIPTION:
The selectin of an embryo for transfer is currently based on detailed morphological assessment and scoring system. morhpokinetics introduced recently to IVF laboratories can define annotations and provide an algorithm for optimal cleavage rates and embryonic development. however more data and validations are requested when it comes to choosing the best single embryo from a cohort of available similarly graded embryos. Consequently, non-invasive quantitative methods for embryo selection prior to transfer have been sought. In the current study metabolic profile of follicular fluid and the embryos produced in IVF procedure will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF procedures at Carmel Medical Center and are able to sign an informed consent form.
* Female patients age 18-45

Exclusion Criteria:

* Women with any malignancy
* Patient's request to be withdrawn from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants are female patients undergoing IVF procedure in the IVF department in Carmel MC
Study Population: Patients undergoing IVF procedures at Carmel Medical Center
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Different markers discriminating the studied groups. | two years
  High correlation between the studied markers and the currently used morphological assessment of the quality of embryos and oocytes will define the potential of the studied markers as a mean for embryo and quality assessment.
  The current study is pioneer in the field of assessment of embryos and follicles and this group of markers have not been studied previously, therefore we prefer not to clarify more details

CONTACTS AND LOCATIONS:
Overall Officials: Martha Direnfeld, Prof., Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No